CLINICAL TRIAL: NCT06672367
Title: Effects of Balance Training with and Without Gaze Stability Exercises on Cognitive Function Balance and Dynamic Postural Stability in Older Adults with Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/43
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Elderly Population; Cognitive Dysfunction
Keywords: Balance training; Gaze stability exercises; Dynamic postural stability; Balance; Cognitive function; Older adults
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: It will involve two groups. Experimental group involves balance training combined with gaze stability exercises for the treatment of mild cognitive impairment and the control group involves only balance training for the treatment of mild cognitive impairment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Balance Training Group (Experimental): It includes participants receiving balance training for mild cognitive impairment.
  Balance training
  Walking on a flat surface at the beginning of each session for 5-10 minutes Perform different static and dynamic balance exercises along with cognitive tasks.
  Static standing with feet together with eyes open and closed Semi-tandem stand and tandem stand Forward and backward weight shift exercises Counting backwards by threes, Naming object or animals, Recalling a short sequence of numbers or words.
  Side stepping, marching, forward and backward walking Hip extension and abduction Cognitive task includes word association or simple math problems. Standing on one leg Relaxation and breathing exercises including deep inhaling and exhaling or walking slowly at the end of each session for 5-10 minutes During training sessions, balance activities and cognitive tasks will be implemented simultaneously.
  Interventions: Procedure: Balance training group
- Balance Training Combined with Gaze Stability Exercises Group (Experimental): It includes participants receiving balance training combined with gaze stability exercises for mild cognitive impairment.
  Balance training
  Walking on a flat surface at the beginning of each session for 5-10 minutes Perform different static and dynamic balance exercises along with cognitive tasks.
  Static standing with feet together with eyes open and closed Semi-tandem stand and tandem stand Forward and backward weight shift exercises Counting backwards by threes, Naming object or animals, Recalling a short sequence of numbers or words.
  Side stepping, marching, forward and backward walking Hip extension and abduction Cognitive task includes word association or simple math problems. Standing on one leg Relaxation and breathing exercises including deep inhaling and exhaling or walking slowly at the end of each session for 5-10 minutes During training sessions, balance activities and cognitive tasks will be implemented simultaneously.
  Gaze stability exercises
  Visual tracking exercise
  Interventions: Procedure: Balance training combined with gaze stability exercises

INTERVENTIONS:
Procedure: Balance training group — It includes participants receiving balance training for mild cognitive impairment.
  Balance training
  Walking on a flat surface at the beginning of each session for 5-10 minutes Perform different static and dynamic balance exercises along with cognitive tasks.
  Static standing with feet together with eyes open and closed Semi-tandem stand and tandem stand Forward and backward weight shift exercises Counting backwards by threes, Naming object or animals, Recalling a short sequence of numbers or words.
  Side stepping, marching, forward and backward walking Hip extension and abduction Cognitive task includes word association or simple math problems. Standing on one leg Relaxation and breathing exercises including deep inhaling and exhaling or walking slowly at the end of each session for 5-10 minutes During training sessions, balance activities and cognitive tasks will be implemented simultaneously.
  Arms: Balance Training Group
Procedure: Balance training combined with gaze stability exercises — It includes participants receiving balance training combined with gaze stability exercises for mild cognitive impairment.
  Balance training
  Walking on a flat surface at the beginning of each session for 5-10 minutes Perform different static and dynamic balance exercises along with cognitive tasks.
  Static standing with feet together with eyes open and closed Semi-tandem stand and tandem stand Forward and backward weight shift exercises Counting backwards by threes, Naming object or animals, Recalling a short sequence of numbers or words.
  Side stepping, marching, forward and backward walking Hip extension and abduction Cognitive task includes word association or simple math problems. Standing on one leg Relaxation and breathing exercises including deep inhaling and exhaling or walking slowly at the end of each session for 5-10 minutes During training sessions, balance activities and cognitive tasks will be implemented simultaneously.
  Gaze stability exercises
  Visual tracking exercises
  Arms: Balance Training Combined with Gaze Stability Exercises Group

SUMMARY:
The study aims to evaluate the effects of balance training, with and without gaze stability exercises, on cognitive function, balance, and postural stability in older adults with mild cognitive impairment (MCI). A randomized controlled trial with 30 participants will be conducted at Fauji Foundation Hospital and Chakwal. Participants will be divided into two groups: one receiving balance training with gaze stability exercises, and the other receiving balance training alone. Baseline, 4-week, and 8-week assessments will measure cognitive function (Montreal Cognitive Assessment), balance (Berg Balance Scale), and mobility (Time Up and Go test). Training will consist of 24 sessions over 8 weeks, with sessions lasting 30-50 minutes.

DETAILED DESCRIPTION:
OBJECTIVES OF STUDY

1. To determine the effects of balance training with and without gaze stability exercises on cognitive function in older adults with mild cognitive impairment.
2. To determine the effects of balance training with and without gaze stability exercises on balance in older adults with mild cognitive impairment.
3. To determine the effects of balance training with and without gaze stability exercises on mobility in older adults with mild cognitive impairment

HYPOTHESIS

ALTERNATE HYPOTHESIS

1. HA- There is a statistically significant difference in effect of balance training with gaze stability exercises in comparison balance training alone on cognitive function in older adults with MCI. (p<0.05)
2. HA- There is a statistically significant difference in effect of balance training with gaze stability exercises in comparison balance training alone on balance in older adults with MCI. (p<0.05)
3. HA- There is a statistically significant difference in effect of balance training with gaze stability exercises in comparison balance training alone on dynamic postural stability in older adults with MCI. (p<0.05)

NULL HYPOTHESIS

1. H0 - There is no statistically significant difference in effect of balance training with gaze stability exercises in comparison balance training alone on cognitive function in older adults with MCI. (p>0.05)
2. H0 - There is no statistically significant difference in effect of balance training with gaze stability exercises in comparison balance training alone on balance in older adults with MCI. (p>0.05)
3. H0 - There is no statistically significant difference in effect of balance training with gaze stability exercises in comparison balance training alone on dynamic postural stability/mobility in older adults with MCI. (p>0.05)

Research Design: Experimental study. Randomized Control Trial

Clinical setting: Chakwal Study duration: 6 months

Data will be collected on Demographics and general information Cognitive function will be assessed with the help of MOCA (Montreal Cognitive Assessment Scale). Balance will be assessed with the help of BBS (Berg Balance Scale). Dynamic postural stability will be assessed with the help of TUG (Time Up and Go test).

SIGNIFICANCE OF STUDY:

Mild Cognitive Impairment (MCI) is a major risk factor for dementia among older adults, although research into its neurological features is limited. Addressing this gap is crucial given the interrelationship of balance issues and cognitive decline. Combining balance training with gaze stability exercises provides a comprehensive intervention method that shows potential for improving both balance and cognitive function. Studies have highlighted the potential benefits of these therapies for improving overall well-being and functional independence in older persons with MCI. Investigating their combined effects provides valuable insights into optimizing rehabilitation strategies for cognitive function, balance, and dynamic postural stability, thereby contributing to improving quality of life and reducing fall risk in this vulnerable population. This research aims to add data to the existing literature

, exploring tailored interventions that address both physical and cognitive aspects simultaneously. By providing understanding on the effectiveness of such interventions, this study seeks to enhance the care and management of older adults with MCI, ultimately promoting better outcomes and quality of life for this population.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 55 years and above older adults.
* Both male and female.
* Having mild cognitive impairment (MCI) having score of 18-25 on Montreal Cognitive Assessment Scale (Urdu version).
* Ability to understand simple instruction and those who are capable of participating in physical exercise programs.

Exclusion Criteria

* Diagnosed neurological and psychiatric disorders.
* Those unable to engage in physical activity due to mobility limitations.
* Individuals with significant visual and hearing impairments affecting participation in gaze stability exercises.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | 8 weeks
  Cognitive function will be assesed by using montreal cognitive assessment scale.
  It has a total score of 30, with higher numbers indicating better Cognition Function. A normal score is regarded to be 26 or higher.
  18-25 = mild cognitive impairment
Balance | 8 weeks
  Balance will be assessed by using berg balance scale. It is a 14-item objective measure. It is a widely used tool for assessing balance in various populations. The scoring system ranges from 0 to 56, where higher scores indicate better balance. Total scores of 0 to 20 indicate a high risk for falls, 21 to 40 indicate a moderate risk, and 41 to 56 indicate a low risk in adults.
Dynamic Postural Stability | 8 weeks
  Dynamic Postural Stability will be assessed by using time up and go test. It assesses mobility, balance, walking ability, and fall risk in older adults. It is administered in less than 3 minutes. Scoring of < 10 seconds is considered normal. As the time duration to complete the test increases the risk of fall increases indicating poor dynamic postural stability and mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan